CLINICAL TRIAL: NCT03054870
Title: A Comparison of Technegas® and Xenon 133 Planar Lung Imaging in Subjects Referred for Ventilation Scintigraphy
Brief Title: A Comparison of Technegas and Xenon-133 Planar Lung Imaging in Subjects Referred for Ventilation Scintigraphy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Trial met primary efficacy endpoint target. No additional subjects necessary.
Sponsor: Cyclomedica Australia PTY Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CYC-009
Record Dates: First submitted 2017-02-08; First posted 2017-02-16 (Actual); Results first posted 2021-09-24 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-08

CONDITIONS: Lung Structure Determination
Keywords: pulmonary ventilation; ventilation scintigraphy
MeSH Terms: interventions — Xenon-133; Lasers, Gas; Technegas

STUDY DESIGN:
Intervention Model Description: Subjects will undergo standard of care Xe-133 ventilation scintigraphy per medical needs followed by investigational Technegas ventilation scintigraphy per protocol.
Masking Description: Independent blinded readers will assess all ventilation scintigraphy images, masked as to subject identity and re-identified with a unique random code number (different code numbers for Xe-133 and Technegas images). The Xe-133 and Technegas images will be read in separate reading sessions in random order.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Xe-133 Followed by Technegas (Other): Subjects first inhaled active comparator Xe-133, approximately 10 to 30 millicuries (mCi), and ventilation planar scintigraphy was performed per site standard of care procedures for subject medical need. On the same day, following completion of Xe-133 imaging, subjects inhaled experimental Technegas (Technetium-99m labeled carbon particles), approximately 1.1 mCi, and ventilation planar scintigraphy was performed.
  Interventions: Drug: Xe-133; Drug: Technegas

INTERVENTIONS:
Drug: Xe-133 — Xe-133 ventilation scintigraphy
  Other Names: Xenon-133; Xenon gas
Drug: Technegas — Technegas ventilation scintigraphy
  Other Names: Technetium-99m labeled carbon particles

SUMMARY:
Phase 3 within-subject non-inferiority trial of Technegas ventilation imaging compared to Xenon-133 (Xe-133) ventilation imaging to demonstrate the non-inferiority of Technegas compared to Xe-133 ventilation studies with respect to subject pulmonary ventilatory distribution. Subjects will undergo site-specific standard of care (SOC) Xe-133 imaging per medical needs followed by Technegas ventilation imaging per study protocol.

DETAILED DESCRIPTION:
This is a Phase 3 within-subject non-inferiority trial of Technegas ventilation imaging compared to Xenon-133 (Xe-133) ventilation imaging to demonstrate the non-inferiority of Technegas compared to Xe-133 ventilation studies with respect to subject pulmonary ventilatory distribution. Subjects will undergo site-specific standard of care (SOC) Xe-133 imaging per medical needs followed by Technegas ventilation imaging per study protocol. Primary assessments of efficacy will be based on three blinded readers' assessments of the Technegas and Xe-133 ventilation images in independent reading sessions.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject at least 18 years of age.
* Subject is a candidate for ventilation imaging.
* Subject must be willing and able to provide informed consent.
* Subject must be stable and able to undergo Xe-133 planar imaging and Technegas planar imaging.
* Subject must be willing and agree to complete study procedures.
* Subject is using adequate birth control, if female and fertile. Adequate birth control is defined as surgical sterilization, hormone contraceptive use or intrauterine device (IUD).
* Female subject of child-bearing potential has a negative urine or serum pregnancy test.
* Subject has had or is scheduled to have a chest X-ray within 24 hours prior to the investigational imaging study.

Exclusion Criteria:

* Subject has been administered any other radiopharmaceutical within a timeframe that might cause interference with study imaging.
* Subject is a pregnant or lactating female.
* Subject has received Technegas in the past.
* Subject has received an investigational drug within 30 days prior to dosing.
* Subject is hemodynamically unstable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-09-18 (Actual); Study Completion 2020-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward M Aten, MD, Study Director — Certus International, Inc.
Locations (9):
- United States (9):
  - Morton Plant Hospital, Clearwater, Florida
  - Mayo Clinic in Jacksonville, FL, Jacksonville, Florida
  - Loyola University Medical Center, Maywood, Illinois
  - Washington University Medical Center, Barnes-Jewish Hospital - Center for Advanced Medicine, St Louis, Missouri
  - Duke University Hospital, Durham, North Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Scott & White Medical Center, Temple, Texas
  - University of Utah Health Science Center, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Day of Ventilation Imaging
Arm/Group | Xe-133 Followed by Technegas
Started | 210 (16 of 226 enrolled subjects were withdrawn from the study prior to receiving Technegas and were not included in further study assessments.)
Completed | 205
Not Completed | 5
Not completed — Protocol Violation | 4
Not completed — Lost to Follow-up | 1
Period: 24-hour Follow-up
Arm/Group | Xe-133 Followed by Technegas
Started | 118 (24-hour follow-up was omitted from Protocol Amendment 1, so 92 subjects enrolled under Amendment 1 not included.)
Completed | 118
Not Completed | 0
Period: Blinded Read of Images
Arm/Group | Xe-133 Followed by Technegas
Started | 200 (At time of study termination, 200 subjects had completed the blinded read assessments. The decision to terminate was based on the positive results of an unplanned interim analysis of these blind read data by a third party statistician.)
Completed | 200
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety cohort - subjects who received any dose of Technegas
Groups:
- Xe-133 Followed by Technegas: Subjects received the active comparator Xe-133 followed by inhalation of experimental Technegas on the same day.
Arm/Group | Xe-133 Followed by Technegas
Number analyzed (Participants) | 210
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (13.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99
  Male | 111
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 205
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 22
  White | 186
  More than one race | 0
  Unknown or Not Reported | 0
Body Mass Index [Mean (Standard Deviation); unit: kilogram/meter squared] — Population: 4 participants had unknown weight or height
  kilogram/meter squared
    number analyzed (Participants) | 206
    (all) | 29.14 (7.472)
Reason for Ventilation Imaging [Count of Participants; unit: Participants] — Subjects could have more than one reason checked for ventilation imaging. Suspected pulmonary embolism (PE) includes subjects presenting with chest pain, shortness of breath or dyspnea.
  In 58 cases pre-lung surgery evaluation was checked in addition to another lung disease category; in 39 cases lung surgery evaluation (pre or post) was the only reason checked.
  Generally, "Other" reason was checked in addition to one of the other specified categories
  Participants
    Suspected Pulmonary Embolism (PE) or Follow-up for PE: Yes | 71
    Suspected Pulmonary Embolism (PE) or Follow-up for PE: No | 139
    Chronic Obstructive Pulmonary Disease (COPD): Yes | 35
    Chronic Obstructive Pulmonary Disease (COPD): No | 175
    Pulmonary or Cystic Fibrosis: Yes | 31
    Pulmonary or Cystic Fibrosis: No | 179
    Pulmonary Hypertension: Yes | 25
    Pulmonary Hypertension: No | 185
    Pre or Post Lung Surgery Evaluation (Lung Transplant or Reduction): Yes | 97
    Pre or Post Lung Surgery Evaluation (Lung Transplant or Reduction): No | 113
    Other Reason: Yes | 37
    Other Reason: No | 173
Screening Chest X-Ray [Count of Participants; unit: Participants] — Screening chest X-ray was performed according to each site's standard of care prior to ventilation imaging.
  Participants
    Interpretation Normal | 67
    Interpretation Abnormal | 143
Pleural Effusion Observed in Screening Chest X-Ray [Count of Participants; unit: Participants]
  Yes | 12
  No | 198

OUTCOME MEASURES:

1. Primary Outcome: Blinded Readers Percent Agreement (PA) for Matching Image Views
Description: Three blinded readers independently assessed the Xe-133 and Technegas images in separate reading sessions. Readers were blinded to all clinical information except a subject's screening chest X-ray. Xe-133 images were obtained per site-specific standard of care. Technegas images included a 6-view image set, and the primary endpoint was based on assessment of the subset of views that matched the Xe-133 image views. At the start of each case-read, a reader visually divided each lung into 3 regions of approximately equal size arranged craniocaudally (apical, mid, and basal), 6 regions in total, and then assessed each lung region for ventilation according to a three-point scale: 0=absent ventilation, 1=decreased ventilation, 2=normal ventilation. At the unplanned interim stage, PA between the Xe-133 scores and Technegas scores was tested for non-inferiority at one-sided alpha=0.0141, equivalent to the lower bound of the 97.18% confidence interval exceeding 60%.
Time Frame: The median duration of Technegas imaging was 22 minutes. Blinded reader assessments of images ranged from <1 month to 16 months following the imaging (median 5 months).
Population: Full Analysis Set (FAS) consisting of subjects who completed all of the ventilation imaging on the study, and both sets of Xe-133 planar scans and the Technegas planar scans were of interpretable image quality according to site Investigators' assessment.
Measure: Number (97.18% Confidence Interval); unit: percentage of lung regions
Groups:
- Blinded Reader 03: Blinded Reader 03's Percent Agreement between Xe-133 and Technegas Ventilation Scores based on Matched image views.
- Blinded Reader 04: Blinded Reader 04's Percent Agreement between Xe-133 and Technegas Ventilation Scores based on Matched image views.
- Blinded Reader 05: Blinded Reader 05's Percent Agreement between Xe-133 and Technegas Ventilation Scores based on Matched image views.
Arm/Group | Blinded Reader 03 | Blinded Reader 04 | Blinded Reader 05
Number analyzed (Participants) | 200 | 200 | 200
percentage of lung regions | 76.2 [72.3 to 79.6] | 70.7 [66.4 to 74.7] | 80.1 [76.4 to 83.3]
Statistical Analysis 1: Comparison: Blinded Reader 03 vs Blinded Reader 04 vs Blinded Reader 05; PA between Technegas and Xe-133 from analysis of each of the 3 blinded readers' ventilation scores was subjected to the following test of null (H0) versus alternate hypotheses (HA): H0: PA <= 60% versus HA: PA > 60%. The original sample size of 240 subjects was based on 90% power and one-sided alpha=0.025. For the unplanned interim analysis of 200 subjects, testing for non-inferiority used one-sided alpha=0.0141 (critical value provided by lower bound of the 97.18% confidence interval); Test type: Non-Inferiority — The non-inferiority margin was determined from a separate study where 6 blinded readers read and re-read 75 Xe-133 planar ventilation imaging studies in 2 read sessions separated by a minimum of 4 weeks. The readers scored the 6 regions of the lung using the same ventilation scoring metric used in this study. Based on analysis of the read/re-read results, 60% was established as a suitable margin for establishing the non-inferiority of Technegas compared to Xe-133; p < 0.0141, Mixed Models Analysis — P-value is one-sided; for testing non-inferiority the associated critical value for PA is provided by lower bound of the 97.18% confidence interval; Binary agreement scores between Technegas and Xe-133 ventilation scores by subject-lung region served as the dependent variable in the model; Binary agreement scores were analyzed for each reader separately using a generalized linear model with SAS® PROC GENMOD. The logit function (log odds ratio) was specified as the link function, and subject was specified as a repeated measure to allow for correlations between lung regions within a subject. The estimate of the intercept of the model using generalized estimating equation (GEE) methodology provided an overall estimate of the agreement and corresponding confidence interval in terms of the log odds ratio. Simple algebra was used to obtain the corresponding estimates and confidence intervals in terms of percent agreement (PA). For the study to be considered a success, the null hypothesis had to be rejected for at least 2 of the 3 blinded readers for the primary efficacy endpoint

2. Secondary Outcome: Blinded Readers Percent Agreement (PA) for All Image Views
Description: Three blinded readers independently assessed the Xe-133 and Technegas images in separate reading sessions. Readers were blinded to all clinical information except a subject's screening chest X-ray. Xe-133 images were obtained per site-specific standard of care. Technegas images included a 6-view image set. Two sequential reads were conducted of each subject's Technegas images. In the first read, only views that matched the Xe-133 image views were presented and read, and assessments based on the matched views were used in the primary outcome measure. Immediately following the commitment of those assessments, all Technegas image views were presented to the reader, and a second assessment of all the Technegas image views was made using the same ventilation scoring metric as described for the primary outcome measure. The estimation of PA and its analyses were also the same as for the primary outcome measure.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (97.18% Confidence Interval); unit: percentage of lung regions
Groups:
- Blinded Reader 03: Blinded Reader 03's Percent Agreement between Xe-133 and Technegas Ventilation Scores based on All image views.
- Blinded Reader 04: Blinded Reader 04's Percent Agreement between Xe-133 and Technegas Ventilation Scores based on All image views.
- Blinded Reader 05: Blinded Reader 05's Percent Agreement between Xe-133 and Technegas Ventilation Scores based on All image views.
Arm/Group | Blinded Reader 03 | Blinded Reader 04 | Blinded Reader 05
Number analyzed (Participants) | 200 | 200 | 200
percentage of lung regions | 75.7 [71.7 to 79.2] | 69.1 [64.7 to 73.2] | 79.6 [75.6 to 83.0]
Statistical Analysis 1: Comparison: Blinded Reader 03 vs Blinded Reader 04 vs Blinded Reader 05; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.0141, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; [other analysis details as in outcome 1, analysis 1]

3. Secondary Outcome: Percent Agreement Measuring Inter-observer Agreement
Description: Percent agreement (PA) measuring inter-observer agreement between pairs of blinded readers for their ventilation scoring assessments within each of the three imaging groups: Xe-133, Technegas matched views, and Technegas all views. For each image set, a reader scored 6 regions of the lungs according to a three-point scale: 0=absent ventilation, 1=decreased ventilation, 2=normal ventilation; agreement between a pair of readers' assessments was based on the agreement of their ventilation scores by subject and lung region.
Time Frame: as for outcome 1
Population: Full Analysis Set (FAS)
Measure: Number (95% Confidence Interval); unit: percentage of lung regions
Groups:
- Xe-133 PA: Percent agreement (PA) between a pair of blinded readers ventilation lung scores based on assessment of Xe-133 image views.
- Technegas PA Matched Views: Percent agreement (PA) between a pair of blinded readers ventilation lung scores based on assessment of Technegas image views that matched the Xe-133 image views.
- Technegas PA All Views: Percent agreement (PA) between a pair of blinded readers ventilation lung scores based on assessment of all Technegas image views.
Arm/Group | Xe-133 PA | Technegas PA Matched Views | Technegas PA All Views
Number analyzed (Participants) | 200 | 200 | 200
percentage of lung regions
  Reader Pair 03, 04 | 82.8 [79.9 to 85.4] | 72.7 [69.0 to 76.1] | 71.6 [67.8 to 75.1]
  Reader Pair 03, 05 | 80.4 [76.9 to 83.5] | 81.2 [78.1 to 84.0] | 80.8 [77.6 to 83.7]
  Reader Pair 04, 05 | 79.6 [76.1 to 82.7] | 73.9 [70.0 to 77.4] | 73.4 [69.4 to 77.1]
Statistical Analysis 1: Comparison: Xe-133 PA vs Technegas PA Matched Views vs Technegas PA All Views; Test type: Other; Estimates of inter-observer percent agreement were obtained as follows. For each reader-pair, binary agreement scores by subject and lung region were analyzed using a generalized linear model with SAS® PROC GENMOD. The logit function (log odds ratio) was specified as the link function, and subject was specified as a repeated measure to allow for correlations between lung regions within a subject. The estimate of the intercept of the model using generalized estimating equation (GEE) methodology provided an overall estimate of the agreement and corresponding confidence interval in terms of the log odds ratio. Simple algebra was used to obtain the corresponding estimates and confidence intervals in terms of percent agreement

4. Secondary Outcome: Kappa Statistics Between Pairs of Blinded Readers by Lung Region
Description: By lung-region kappa statistics measuring inter-observer agreement between pairs of blinded readers for their ventilation scoring assessments within each of the three imaging groups: Xe-133, Technegas matched views, and Technegas all views. For each image set, a reader scored 6 regions of the lungs according to a three-point scale: 0=absent ventilation, 1=decreased ventilation, 2=normal ventilation. Kappa statistics for a pair of readers' assessments were derived from the frequencies of the cross-tabulation of the readers' ventilation scores by lung region. Kappa statistics are an index of inter-observer agreement corrected for chance with possible values ranging from -1 to 1, where 1 represents perfect agreement.
Time Frame: as for outcome 1
Population: Full Analysis Set (FAS)
Measure: Number (95% Confidence Interval); unit: Index of inter-reader agreement
Groups:
- Xe-133 Kappa: Kappa statistics for a pair of blinded readers ventilation lung scores based on assessment of Xe-133 image views.
- Technegas Kappa Matched Views: Kappa statistics for a pair of blinded readers ventilation lung scores based on assessment of Technegas image views that matched the Xe-133 image views.
- Technegas Kappa All Views: Kappa statistics for a pair of blinded readers ventilation lung scores based on assessment of all Technegas image views.
Arm/Group | Xe-133 Kappa | Technegas Kappa Matched Views | Technegas Kappa All Views
Number analyzed (Participants) | 200 | 200 | 200
Index of inter-reader agreement
  Left Lung Apical: Pair 03, 04 | 0.479 [0.339 to 0.619] | 0.529 [0.428 to 0.630] | 0.503 [0.404 to 0.602]
  Left Lung Apical: Pair 03, 05 | 0.500 [0.365 to 0.634] | 0.558 [0.446 to 0.670] | 0.589 [0.479 to 0.700]
  Left Lung Apical: Pair 04, 05 | 0.538 [0.406 to 0.671] | 0.481 [0.369 to 0.592] | 0.467 [0.360 to 0.573]
  Left Lung Mid: Pair 03, 04 | 0.551 [0.423 to 0.680] | 0.474 [0.371 to 0.577] | 0.509 [0.405 to 0.612]
  Left Lung Mid: Pair 03, 05 | 0.538 [0.408 to 0.669] | 0.560 [0.440 to 0.681] | 0.571 [0.457 to 0.685]
  Left Lung Mid: Pair 04, 05 | 0.527 [0.401 to 0.653] | 0.434 [0.332 to 0.535] | 0.421 [0.320 to 0.521]
  Left Lung Basal: Pair 03, 04 | 0.530 [0.416 to 0.644] | 0.466 [0.368 to 0.563] | 0.452 [0.355 to 0.549]
  Left Lung Basal: Pair 03, 05 | 0.517 [0.401 to 0.633] | 0.553 [0.445 to 0.662] | 0.510 [0.399 to 0.621]
  Left Lung Basal: Pair 04, 05 | 0.469 [0.350 to 0.588] | 0.424 [0.321 to 0.528] | 0.461 [0.359 to 0.564]
  Right Lung Apical: Pair 03, 04 | 0.665 [0.535 to 0.795] | 0.484 [0.389 to 0.580] | 0.495 [0.400 to 0.591]
  Right Lung Apical: Pair 03, 05 | 0.589 [0.464 to 0.713] | 0.621 [0.512 to 0.730] | 0.596 [0.484 to 0.708]
  Right Lung Apical: Pair 04, 05 | 0.581 [0.452 to 0.710] | 0.593 [0.490 to 0.696] | 0.559 [0.459 to 0.660]
  Right Lung Mid: 03, 04 | 0.583 [0.445 to 0.721] | 0.518 [0.412 to 0.624] | 0.464 [0.357 to 0.571]
  Right Lung Mid: 03, 05 | 0.478 [0.348 to 0.607] | 0.663 [0.554 to 0.772] | 0.682 [0.578 to 0.786]
  Right Lung Mid: 04, 05 | 0.511 [0.380 to 0.642] | 0.530 [0.426 to 0.634] | 0.515 [0.410 to 0.619]
  Right Lung Basal: 03, 04 | 0.486 [0.367 to 0.605] | 0.448 [0.353 to 0.543] | 0.427 [0.333 to 0.521]
  Right Lung Basal: 03, 05 | 0.479 [0.360 to 0.597] | 0.530 [0.418 to 0.642] | 0.533 [0.424 to 0.642]
  Right Lung Basal: 04, 05 | 0.519 [0.403 to 0.634] | 0.496 [0.395 to 0.597] | 0.509 [0.406 to 0.611]
Statistical Analysis 1: Comparison: Xe-133 Kappa vs Technegas Kappa Matched Views vs Technegas Kappa All Views; Test type: Other; For each pair of readers, by lung region estimates of kappa statistics and their corresponding 95% confidence intervals were generated from cross-tabulation frequencies of the readers' ventilation scores using SAS® PROC FREQ and the AGREE option

ADVERSE EVENTS:
Time Frame: From the time of Informed Consent until study discharge. Under the original protocol discharge followed 24-hour follow-up. Under the amended protocol, 24-hour follow-up was removed and discharge followed study imaging.
Arm/Group | Xe-133 Followed by Technegas
All-Cause Mortality (participants affected / at risk) | 0/210
Serious Adverse Events (participants affected / at risk) | 0/210
Other Adverse Events (participants affected / at risk) | 7/210
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Xe-133 Followed by Technegas (N=210)
Dizziness (Nervous system disorders) | 2 (2)
Dysgeusia (Nervous system disorders) | 2 (2)
Chills (General disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Unblinded analysis of imaging efficacy data was to be done at completion of study and all blinded readings. Due to the COVID-19 pandemic impact on enrollment, FDA recommended an unplanned interim analysis be performed using blind read data from 200 subjects. Interim analysis was done by independent 3rd party statistician and reviewed by a Data Efficacy Monitoring Committee (DEMC), which recommended termination of the study based on positive results. Sponsor agreed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan: Original Prototocol (2016-10-04): https://cdn.clinicaltrials.gov/large-docs/70/NCT03054870/Prot_SAP_000.pdf
  • Study Protocol and Statistical Analysis Plan: Protocol Amendment 1 (2018-11-02): https://cdn.clinicaltrials.gov/large-docs/70/NCT03054870/Prot_SAP_001.pdf
  • Statistical Analysis Plan: Addendum for Statistical Analysis Plan (2020-07-30): https://cdn.clinicaltrials.gov/large-docs/70/NCT03054870/SAP_002.pdf